CLINICAL TRIAL: NCT05899205
Title: Patient Recorded Indexing Measurements
Acronym: PRIMs
Status: Recruiting | Type: Observational
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: Zuyderland Medisch Centrum (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Nicole Hildebrand, Coordinating Investigator, Academisch Ziekenhuis Maastricht
Other Study IDs: NL65402.068.18
Record Dates: First submitted 2023-02-16; First posted 2023-06-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cachexia; Cancer; Weight, Body
Keywords: Cancer cachexia; Physical activity; Body weight; Body composition; Functional mobility; Pre-treatment assessment
MeSH Terms: conditions — Cachexia; Neoplasms; Body Weight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be freezed at -80°C and will be stored for 15 years and analyzed if new insights related to this research should arise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Periampullary and pancreatic cancer: Patients undergoing curative-intent treatment for periampullary or pancreatic cancer.
- Upper-GI Cancer: Patients undergoing curative-intent treatment for esophageal or gastric cancer
- Lower-GI Cancer: Patients undergoing curative-intent treatment for colorectal cancer or colorectal liver metastases
- Hepatic cancer: Patients undergoing curative-intent treatment for hepatocellular carcinoma or intrahepatic or perihilar cholangiocarcinoma
- Gynecological cancer: Patients undergoing curative-intent treatment for ovarian, cervical, and endometrial cancer

SUMMARY:
Rationale: One of the greatest challenges in the field of cancer treatment is cachexia, a multifactorial syndrome characterized by substantial loss of body weight (muscle and fat mass), leading to progressive functional impairment. Cancer cachexia significantly impairs quality of life and survival as well as treatment outcome. Despite its considerable relevance for the prognosis of cancer patients, the diagnosis of cachexia is problematic. The current consensus definition of cancer cachexia is based on weight loss over the last six months. In practice, this is assessed by subjective reporting by the patient, which is subject to error and bias. Novel technologies enable accurate, standardized, and objective assessment of body weight and physical activity by newly diagnosed cancer patients in the home situation. Because of the increasing implementation of neo-adjuvant treatment strategies that offer an extended time-window for the collection of these data, there is a great opportunity to use this information in risk analyses by treating physicians, optimization of pre-habilitation programs, and in the shared-decision making process with the patient.

Objective: The central aim of the 'Patient-Recorded Indexing MeasurementS' (PRIMS) study is to improve the accuracy of the diagnosis of cachexia in patients with cancer. This aim will be achieved by focusing on two objectives. The primary objectives are to compare self-reported and objectively measured pre-treatment weight change. The secondary objectives are to define host phenotypes and to investigate longitudinal associations between body weight and physical activity patterns.

Study design: Explorative pilot study

Study population: Patients ≥18 years old undergoing curative-intent chemotherapy or surgery for cancer. Patients will be included in two referral centers specialized in treatment of patients with upper gastrointestinal, hepatobiliary, pancreatic, colorectal, and ovarian cancer.

Main study parameters/endpoints: The primary endpoint is body weight change over time. Objectively measured body weight will be compared to subjectively reported body weight change. Their respective association with treatment-related adverse events and survival will be investigated. Survival will be calculated from date of start of treatment until death. Chemotherapy related adverse event will be recorded using the Common Terminology Criteria for Adverse Events. Postoperative adverse events will be scored according to the Clavien-Dindo classification.

Secondary endpoints: The secondary endpoints will be the association between other cachexia-related parameters that are investigated in the study and adverse events / survival. Other parameters include physical activity over time, using accelerometry, baseline physical assessment, anthropometric measurements, body composition, and laboratory results. Besides this, other endpoints that will be assessed are disease-free survival (calculated from the first day of treatment until first recurrence) and response to chemotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

DETAILED DESCRIPTION:
Patients undergoing curative-intent chemotherapy or surgery for cancer will be included. All types of cancer might be included. To date, the two participating centers are referral hospitals focused on the care of hepatobiliary, pancreatic, upper-GI, colorectal, and ovarian cancer.

Upon informed consent, patients will undergo extensive pre-treatment screening. The screening consists of physical assessment and anthropometric measurements. The physical assessment consists of a modified steep-ramp test, 30-second chair stand test, handgrip strength, timed-up-and-go-test, and 2-minute walk test. For anthropometric measurements the study personnel will measure current BMI (kg/m^2), waist circumference (cm), upper arm circumference (cm), triceps skinfold (mm), and wrist circumference (cm). Upper arm muscle and fat area (cm^2) will be calculated based on triceps skinfold and upper arm circumference.

All measurements will be performed by a trained physiotherapist or nurse practitioner, if available. The study team will also be trained to perform measurements.

Moreover, body composition will be measured at baseline and after treatment. Body composition will be assessed at the level of the third lumbar level (L3) where both processi transversi are visible. Body composition analysis will be performed using an automated segmentation algorithm (MosaMatic (TM) ). The assessed areas are skeletal muscle, visceral adipose tissue, and subcutaneous adipose tissue. For each area indices (cm^2/m^2) corrected for body length and radiation attenuation (HU) will be measured.

Laboratory results include, but are not limited to, C-reactive protein (CRP) (mg/L), lymphocyte count, albumin (g/L), HbA1c, haemoglobin, CRP, TNF-α, interleukin-6, blood lipids, and additional parameters related to inflammation

Then, patients receive a weight scale for daily at-home measurements of body weight and an accelerometer for assessing physical activity. Body weight data will be collected using an electronic weight scale with integrated memory SD cards for automated autonomous storage of data (CE licensed). Physical activity will be monitored through a research grade wrist-worn accelerometer that records movement in three axes as well as body position (sedentary versus standing position). Data on frequency, intensity, and duration of activity will be collected. Activity can be summarized into light, moderate and (very) vigorous activity. Additionally, data on sedentary behavior will be collected.

Monitoring plan for patients treated with chemotherapy:

T0 Start of monitoring: When patients first present at the outpatient clinic, they will receive extensive physical analysis as described above. Additionally, the investigators will collect one blood sample. Patients will receive equipment (weight scale and accelerometer) for at home monitoring. The patient will start using the weight scale daily and wear the accelerometer continuously after screening.

T1: Start of chemotherapy: During chemotherapy, the body weight and physical activity measurements will continue. Patients will use the scale once daily and the accelerometer continuously.

T2: End of chemotherapy: The monitoring will continue until two weeks after chemotherapy.

T3: End of monitoring ( usually 2-3 weeks after completion of chemotherapy). A routine CT-scan to assess the effect of the chemotherapy will be performed. Patients will hand in all equipment to the researcher during regular follow-up.

Body composition measurement on the diagnostic CT-scan will be repeated, as described above.

Monitoring plan for patients treated with surgery:

T0 start of monitoring: When patients first present at the outpatient clinic, they will receive extensive physical analysis as described above. Additionally, the investigators will collect one blood sample. Patients will receive equipment (weight scale and accelerometer) for at home monitoring. The patient will start using the weight scale daily and wear the accelerometer continuously.

T1: Hospital admission:

At the day of admission, the patient will not bring the weight scale and accelerometer to the hospital. Monitoring will be paused for the length of hospital stay for primary surgery.

T2: Discharge from hospital:

At the day of discharge after primary surgery, length of stay at the hospital will be recorded. The patient will be reminded to restart monitoring and use the weight scale daily and wear the accelerometer continuously.

T3: End of monitoring:

During the regular follow-up visit 2-3 weeks after discharge, monitoring will end. Patients will hand in all equipment to the researcher during the regular follow-up visit. Over the course of the oncological follow-up, a routine CT-scan will be performed. Body composition analysis at the L3-level will be repeated as described above.

Outcome measurements:

Outcome measurements are presented in their order of registry.

The first outcome measurement is treatment-related adverse events. During chemotherapy adverse events will be recorded according to the Common Toxicity Criteria version 5.0 (www.eortc.be/services/doc/ctc/). For each adverse event the respective number of cycle, type of adverse event, and grade thereof will be recorded. Moreover, for chemotherapy delay, reason for delay, and dose reduction (including %of dose reduction of the respective drug) will be recorded.

Adverse events after surgery will be recording using the Clavien-Dindo classification up to 30 days after surgery. For each complication, the Clavien-Dindo grade will be recorded. Major complications are defined as ≥III.

Averse events will be recorded by a trained physician.

Treatment response after treatment will be graded based on Response Evaluation Criteria in Solid Tumor (RECIST) after chemotherapy. RECIST-criteria will be scored as 'complete response' , 'partial response', 'stable disease', and 'progressive disease'. The criteria will be scored by the radiologist according to international criteria.

Moreover, pathological outcomes will be recorded for solid tumor using the TNM-classification. This includes the extent of the tumor (T), extent of spread to lymph nodes (N), number of resected lymph nodes and number of positive lymph nodes, metastatic disease (M), resection margin (R), perineural invasion, and vascular invasion. The pathological analysis will be performed according to national guidelines.

Survival and disease-free survival will also be recorded. The follow-up will continue up to five years after the last treatment.

Survival will be calculated from the first day of treatment until death. If available, reason of death will also be recorded.

Disease-free survival is defined from the first day of treatment until first sign of recurrence.

Sample size calculation The sample size calculation was based on the primary objective, which is to assess the agreement of cancer cachexia diagnosis based on self-reported weight loss versus objectively measured weight loss. Assuming a null hypothesis intraclass correlation coefficient (ICC) of 0.75, based on previously published literature, and an expected ICC of 0.65, with a significance level of 0.05 and statistical power of 90%, 270 subjects will be required. With an expected dropout rate of 10%, the total sample size is 300.

Data analysis plan Data analysis will be performed using R in the latest version available at the time of analysis (R Foundation for Statistical Computing, Vienna, Austria).

A short data analysis plan is presented here. For the primary objectives of the study, namely, to detect the agreement of cancer cachexia diagnosis based on self-reported weight versus objectively measured body weight and their respective association with treatment-related adverse events and treatment outcomes, the subjective self-reported weight change over the last six months and objective body weight data before treatment from the digital body weight scale will be used. The association between predictive variables and the occurrence of adverse events will be investigated through univariable and multivariable logistic regression analysis.

Predictive parameters include baseline measurements, body composition measurements, and physical activity. Moreover, the correlation between self-reported pre-treatment weight changes versus objectively measured weight changes will be evaluated.

Dissemination policy Research results, negative or positive, will be submitted for publication in peer-reviewed scientific journals. A writing committee, assigned by the principal investigators, will prepare the manuscripts. Co-authorship is reserved for all who contributed constructively to the study at the discretion of the principal investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosed with cancer
* Planned for curative-intent surgery or neo-adjuvant chemotherapy

Exclusion Criteria:

* ASA-classification V,
* severe liver cirrhosis Child grade C,
* end stage renal disease requiring dialysis,
* severe heart disease New York Heart Association class IV,
* chronic obstructive pulmonary disease (COPD) requiring (home)oxygen therapy,
* Patients must be "mobile". They may not be bedridden or in a wheelchair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, requiring neo-adjuvant chemotherapy or curative-intent surgery for cancer
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | throughout treatment, average of 5-14 weeks
  At home measurement with memory integrated weight scale
Number of treatment-related adverse events as assessed by CTCAE v5.0 | throughout treatment, average of 5-14 weeks
  Chemotoxicity according to Common Toxicity Criteria v5.0
Postoperative complications | 30 days postoperatively
  Postoperative complications rated according to Clavien-Dindo classification

SECONDARY OUTCOMES:
Functional mobility/muscle strength | 2-4 weeks before treatment start
  Timed up and go test (in sec)
Functional mobility | 2-4 weeks before treatment start
  2 minute walking test (in m)
Change in body composition (adipose tissue surface and muscular tissue surface) | throughout treatment, average of 5-14 weeks
  Automated segmentation of body composition on the L3 level of abdominal CT-scans
Treatment outcome | after completion of chemotherapy, 5-14 weeks after start of treatment
  Treatment outcome will be evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST)
Physical activity | throughout treatment, average of 5-14 weeks
  Accelerometry data on three axes
Muscle strength | 2-4 weeks before treatment start
  Grip strength analysis (in kg)
Aerobic capacity | 2-4 weeks before treatment start
  Steep ramp test (in W)
Nutritional status | 2-4 weeks before treatment start
  Weight loss before diagnosis
Overall survival | Up to 5 years after completion
  Overall and recurrence free survival
Recurrence free survival | Up to 5 years after completion
  Recurrence free survival

CONTACTS AND LOCATIONS:
Overall Officials: Steven Olde Damink, PhD, MSc., M.D., Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center+, Maastricht
  - Zuyderland Medical Center, Sittard

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perry GS, Byers TE, Mokdad AH, Serdula MK, Williamson DF. The validity of self-reports of past body weights by U.S. adults. Epidemiology. 1995 Jan;6(1):61-6. doi: 10.1097/00001648-199501000-00012. PMID 7888448
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Baracos VE, Martin L, Korc M, Guttridge DC, Fearon KCH. Cancer-associated cachexia. Nat Rev Dis Primers. 2018 Jan 18;4:17105. doi: 10.1038/nrdp.2017.105. PMID 29345251
- [Background] van Dijk DPJ, Krill M, Farshidfar F, Li T, Rensen SS, Olde Damink SWM, Dixon E, Sutherland FR, Ball CG, Mazurak VC, Baracos VE, Bathe OF. Host phenotype is associated with reduced survival independent of tumour biology in patients with colorectal liver metastases. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):123-130. doi: 10.1002/jcsm.12358. Epub 2018 Oct 31. PMID 30378742
- [Background] van Dijk DPJ, Bakers FCH, Sanduleanu S, Vaes RDW, Rensen SS, Dejong CHC, Beets-Tan RGH, Olde Damink SWM. Myosteatosis predicts survival after surgery for periampullary cancer: a novel method using MRI. HPB (Oxford). 2018 Aug;20(8):715-720. doi: 10.1016/j.hpb.2018.02.378. Epub 2018 Mar 5. PMID 29519644
- [Background] van Dijk DP, Bakens MJ, Coolsen MM, Rensen SS, van Dam RM, Bours MJ, Weijenberg MP, Dejong CH, Olde Damink SW. Low skeletal muscle radiation attenuation and visceral adiposity are associated with overall survival and surgical site infections in patients with pancreatic cancer. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):317-326. doi: 10.1002/jcsm.12155. Epub 2016 Oct 26. PMID 27897432
- [Background] Wallengren O, Lundholm K, Bosaeus I. Diagnostic criteria of cancer cachexia: relation to quality of life, exercise capacity and survival in unselected palliative care patients. Support Care Cancer. 2013 Jun;21(6):1569-77. doi: 10.1007/s00520-012-1697-z. Epub 2013 Jan 13. PMID 23314651
- [Background] Ross PJ, Ashley S, Norton A, Priest K, Waters JS, Eisen T, Smith IE, O'Brien ME. Do patients with weight loss have a worse outcome when undergoing chemotherapy for lung cancers? Br J Cancer. 2004 May 17;90(10):1905-11. doi: 10.1038/sj.bjc.6601781. PMID 15138470
- [Background] Cawley J, Maclean JC, Hammer M, Wintfeld N. Reporting error in weight and its implications for bias in economic models. Econ Hum Biol. 2015 Dec;19:27-44. doi: 10.1016/j.ehb.2015.07.001. Epub 2015 Jul 23. PMID 26256130
- [Background] Connor Gorber S, Tremblay M, Moher D, Gorber B. A comparison of direct vs. self-report measures for assessing height, weight and body mass index: a systematic review. Obes Rev. 2007 Jul;8(4):307-26. doi: 10.1111/j.1467-789X.2007.00347.x. PMID 17578381
- [Background] Peddle-McIntyre CJ, Cavalheri V, Boyle T, McVeigh JA, Jeffery E, Lynch BM, Vallance JK. A Review of Accelerometer-based Activity Monitoring in Cancer Survivorship Research. Med Sci Sports Exerc. 2018 Sep;50(9):1790-1801. doi: 10.1249/MSS.0000000000001644. PMID 29683922
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Fearon K, Arends J, Baracos V. Understanding the mechanisms and treatment options in cancer cachexia. Nat Rev Clin Oncol. 2013 Feb;10(2):90-9. doi: 10.1038/nrclinonc.2012.209. Epub 2012 Dec 4. PMID 23207794
- [Background] Sikkens EC, Cahen DL, de Wit J, Looman CW, van Eijck C, Bruno MJ. A prospective assessment of the natural course of the exocrine pancreatic function in patients with a pancreatic head tumor. J Clin Gastroenterol. 2014 May-Jun;48(5):e43-6. doi: 10.1097/MCG.0b013e31829f56e7. PMID 24717227
- [Background] Shintakuya R, Uemura K, Murakami Y, Kondo N, Nakagawa N, Urabe K, Okano K, Awai K, Higaki T, Sueda T. Sarcopenia is closely associated with pancreatic exocrine insufficiency in patients with pancreatic disease. Pancreatology. 2017 Jan-Feb;17(1):70-75. doi: 10.1016/j.pan.2016.10.005. Epub 2016 Oct 11. PMID 27743711
- [Background] Del Fabbro E. Current and future care of patients with the cancer anorexia-cachexia syndrome. Am Soc Clin Oncol Educ Book. 2015:e229-37. doi: 10.14694/EdBook_AM.2015.35.e229. PMID 25993178
- [Background] Bosaeus I. Nutritional support in multimodal therapy for cancer cachexia. Support Care Cancer. 2008 May;16(5):447-51. doi: 10.1007/s00520-007-0388-7. Epub 2008 Jan 15. PMID 18196284
- [Background] Rutten IJ, van Dijk DP, Kruitwagen RF, Beets-Tan RG, Olde Damink SW, van Gorp T. Loss of skeletal muscle during neoadjuvant chemotherapy is related to decreased survival in ovarian cancer patients. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):458-66. doi: 10.1002/jcsm.12107. Epub 2016 Mar 7. PMID 27030813
- [Background] Ozola Zalite I, Zykus R, Francisco Gonzalez M, Saygili F, Pukitis A, Gaujoux S, Charnley RM, Lyadov V. Influence of cachexia and sarcopenia on survival in pancreatic ductal adenocarcinoma: a systematic review. Pancreatology. 2015 Jan-Feb;15(1):19-24. doi: 10.1016/j.pan.2014.11.006. Epub 2014 Dec 4. PMID 25524484
- [Background] Ninomiya G, Fujii T, Yamada S, Yabusaki N, Suzuki K, Iwata N, Kanda M, Hayashi M, Tanaka C, Nakayama G, Sugimoto H, Koike M, Fujiwara M, Kodera Y. Clinical impact of sarcopenia on prognosis in pancreatic ductal adenocarcinoma: A retrospective cohort study. Int J Surg. 2017 Mar;39:45-51. doi: 10.1016/j.ijsu.2017.01.075. Epub 2017 Jan 18. PMID 28110029
- [Background] Peng P, Hyder O, Firoozmand A, Kneuertz P, Schulick RD, Huang D, Makary M, Hirose K, Edil B, Choti MA, Herman J, Cameron JL, Wolfgang CL, Pawlik TM. Impact of sarcopenia on outcomes following resection of pancreatic adenocarcinoma. J Gastrointest Surg. 2012 Aug;16(8):1478-86. doi: 10.1007/s11605-012-1923-5. Epub 2012 Jun 13. PMID 22692586
- [Background] Cooper AB, Slack R, Fogelman D, Holmes HM, Petzel M, Parker N, Balachandran A, Garg N, Ngo-Huang A, Varadhachary G, Evans DB, Lee JE, Aloia T, Conrad C, Vauthey JN, Fleming JB, Katz MH. Characterization of Anthropometric Changes that Occur During Neoadjuvant Therapy for Potentially Resectable Pancreatic Cancer. Ann Surg Oncol. 2015 Jul;22(7):2416-23. doi: 10.1245/s10434-014-4285-2. Epub 2014 Dec 18. PMID 25519927
- [Background] Harimoto N, Shirabe K, Yamashita YI, Ikegami T, Yoshizumi T, Soejima Y, Ikeda T, Maehara Y, Nishie A, Yamanaka T. Sarcopenia as a predictor of prognosis in patients following hepatectomy for hepatocellular carcinoma. Br J Surg. 2013 Oct;100(11):1523-30. doi: 10.1002/bjs.9258. PMID 24037576
- [Background] Huang DD, Wang SL, Zhuang CL, Zheng BS, Lu JX, Chen FF, Zhou CJ, Shen X, Yu Z. Sarcopenia, as defined by low muscle mass, strength and physical performance, predicts complications after surgery for colorectal cancer. Colorectal Dis. 2015 Nov;17(11):O256-64. doi: 10.1111/codi.13067. PMID 26194849
- [Background] Wang SL, Zhuang CL, Huang DD, Pang WY, Lou N, Chen FF, Zhou CJ, Shen X, Yu Z. Sarcopenia Adversely Impacts Postoperative Clinical Outcomes Following Gastrectomy in Patients with Gastric Cancer: A Prospective Study. Ann Surg Oncol. 2016 Feb;23(2):556-64. doi: 10.1245/s10434-015-4887-3. Epub 2015 Dec 14. PMID 26668085
- [Background] Sharma P, Zargar-Shoshtari K, Caracciolo JT, Fishman M, Poch MA, Pow-Sang J, Sexton WJ, Spiess PE. Sarcopenia as a predictor of overall survival after cytoreductive nephrectomy for metastatic renal cell carcinoma. Urol Oncol. 2015 Aug;33(8):339.e17-23. doi: 10.1016/j.urolonc.2015.01.011. Epub 2015 Jun 18. PMID 26094169
- [Background] Yip C, Goh V, Davies A, Gossage J, Mitchell-Hay R, Hynes O, Maisey N, Ross P, Gaya A, Landau DB, Cook GJ, Griffin N, Mason R. Assessment of sarcopenia and changes in body composition after neoadjuvant chemotherapy and associations with clinical outcomes in oesophageal cancer. Eur Radiol. 2014 May;24(5):998-1005. doi: 10.1007/s00330-014-3110-4. Epub 2014 Feb 18. PMID 24535076
- [Background] Prado CM, Baracos VE, McCargar LJ, Reiman T, Mourtzakis M, Tonkin K, Mackey JR, Koski S, Pituskin E, Sawyer MB. Sarcopenia as a determinant of chemotherapy toxicity and time to tumor progression in metastatic breast cancer patients receiving capecitabine treatment. Clin Cancer Res. 2009 Apr 15;15(8):2920-6. doi: 10.1158/1078-0432.CCR-08-2242. Epub 2009 Apr 7. PMID 19351764
- [Background] West MA, van Dijk DPJ, Gleadowe F, Reeves T, Primrose JN, Abu Hilal M, Edwards MR, Jack S, Rensen SSS, Grocott MPW, Levett DZH, Olde Damink SWM. Myosteatosis is associated with poor physical fitness in patients undergoing hepatopancreatobiliary surgery. J Cachexia Sarcopenia Muscle. 2019 Aug;10(4):860-871. doi: 10.1002/jcsm.12433. Epub 2019 May 21. PMID 31115169
- [Background] Kurk S, Peeters P, Stellato R, Dorresteijn B, de Jong P, Jourdan M, Creemers GJ, Erdkamp F, de Jongh F, Kint P, Simkens L, Tanis B, Tjin-A-Ton M, Van Der Velden A, Punt C, Koopman M, May A. Skeletal muscle mass loss and dose-limiting toxicities in metastatic colorectal cancer patients. J Cachexia Sarcopenia Muscle. 2019 Aug;10(4):803-813. doi: 10.1002/jcsm.12436. Epub 2019 May 15. PMID 31094083
- [Background] Sealy MJ, Dechaphunkul T, van der Schans CP, Krijnen WP, Roodenburg JLN, Walker J, Jager-Wittenaar H, Baracos VE. Low muscle mass is associated with early termination of chemotherapy related to toxicity in patients with head and neck cancer. Clin Nutr. 2020 Feb;39(2):501-509. doi: 10.1016/j.clnu.2019.02.029. Epub 2019 Feb 22. PMID 30846324
- [Background] Ryan AM, Prado CM, Sullivan ES, Power DG, Daly LE. Effects of weight loss and sarcopenia on response to chemotherapy, quality of life, and survival. Nutrition. 2019 Nov-Dec;67-68:110539. doi: 10.1016/j.nut.2019.06.020. Epub 2019 Jun 28. PMID 31522087
- [Background] McTiernan A, Friedenreich CM, Katzmarzyk PT, Powell KE, Macko R, Buchner D, Pescatello LS, Bloodgood B, Tennant B, Vaux-Bjerke A, George SM, Troiano RP, Piercy KL; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity in Cancer Prevention and Survival: A Systematic Review. Med Sci Sports Exerc. 2019 Jun;51(6):1252-1261. doi: 10.1249/MSS.0000000000001937. PMID 31095082
- [Background] Hsueh HY, Pita-Grisanti V, Gumpper-Fedus K, Lahooti A, Chavez-Tomar M, Schadler K, Cruz-Monserrate Z. A review of physical activity in pancreatic ductal adenocarcinoma: Epidemiology, intervention, animal models, and clinical trials. Pancreatology. 2022 Jan;22(1):98-111. doi: 10.1016/j.pan.2021.10.004. Epub 2021 Oct 26. PMID 34750076
- [Background] Latrille M, Buchs NC, Ris F, Koessler T. Physical activity programmes for patients undergoing neo-adjuvant chemoradiotherapy for rectal cancer: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Dec 23;100(51):e27754. doi: 10.1097/MD.0000000000027754. PMID 34941028
- [Background] Lugo D, Pulido AL, Mihos CG, Issa O, Cusnir M, Horvath SA, Lin J, Santana O. The effects of physical activity on cancer prevention, treatment and prognosis: A review of the literature. Complement Ther Med. 2019 Jun;44:9-13. doi: 10.1016/j.ctim.2019.03.013. Epub 2019 Mar 20. PMID 31126580
- [Background] Prince SA, Adamo KB, Hamel ME, Hardt J, Connor Gorber S, Tremblay M. A comparison of direct versus self-report measures for assessing physical activity in adults: a systematic review. Int J Behav Nutr Phys Act. 2008 Nov 6;5:56. doi: 10.1186/1479-5868-5-56. PMID 18990237
- [Background] Boyle T, Lynch BM, Courneya KS, Vallance JK. Agreement between accelerometer-assessed and self-reported physical activity and sedentary time in colon cancer survivors. Support Care Cancer. 2015 Apr;23(4):1121-6. doi: 10.1007/s00520-014-2453-3. Epub 2014 Oct 11. PMID 25301224
- [Background] Broderick JM, Ryan J, O'Donnell DM, Hussey J. A guide to assessing physical activity using accelerometry in cancer patients. Support Care Cancer. 2014 Apr;22(4):1121-30. doi: 10.1007/s00520-013-2102-2. Epub 2014 Jan 4. PMID 24389829
- [Background] Delisle Nystrom C, Pomeroy J, Henriksson P, Forsum E, Ortega FB, Maddison R, Migueles JH, Lof M. Evaluation of the wrist-worn ActiGraph wGT3x-BT for estimating activity energy expenditure in preschool children. Eur J Clin Nutr. 2017 Oct;71(10):1212-1217. doi: 10.1038/ejcn.2017.114. Epub 2017 Jul 26. PMID 28745334
- [Derived] Hildebrand ND, Sier MAT, van Kuijk SMJ, Hoeijmakers LSM, Ackermans LLGC, Ubachs J, Stassen L, Ruber NFM, Schaghen-D'Antonio V, Goedegebuure EP, Baade-Corpelijn L, Bongers BC, Stoot J, Sosef M, Lambrechts S, de Vos van Steenwijk PJ, Engelen M, Lubbers T, Blokhuis TJ, Ten Bosch JA, Valkenburg-van Iersel L, de Vos-Geelen J, den Dulk M, van Dijk DPJ, Olde Damink SWM, Rensen SSM. Patient-recorded indexing measurements (PRIMS) - study protocol of a prospective observational cohort study to improve the accuracy of the diagnosis of cancer cachexia. BMC Cancer. 2025 Oct 14;25(1):1572. doi: 10.1186/s12885-025-14979-z. PMID 41087985